CLINICAL TRIAL: NCT06338462
Title: Mobile Health and Oral Testing to Optimize Tuberculosis Contact Tracing in Colombia
Brief Title: Cali Sin Tos Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000034128; R21AI174129 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: target sample size is an anticipated 120 index persons with TB enrolled over three design cycles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Health and Oral Testing (Experimental): to adapt an automated conversation agent (Chatbot) and oral testing as a novel multi-component strategy for implementing TB contact investigation over three phases of participatory co-design
  Interventions: Device: Chatbot; Diagnostic Test: Oral testing

INTERVENTIONS:
Device: Chatbot — The chatbot is a WhatsApp-based, artificial-intelligence powered customer service agent adapted for TB outreach. The objective of the Chatbot is to facilitate information gathering, education, and support throughout TB contact evaluation, ensuring accessible assistance on-demand during and after contact tracing procedures. It operates in a secure data environment that includes end-to-end encryption and has been reviewed and approved by the data protection team within the information technology unit at the Cali Secretariat of Public Health (SoPH) for the study purposes.
Diagnostic Test: Oral testing — Oral testing involves collection of a saliva sample or use of a nylon swab to collect material from the tongue and oral mucosa that is then tested with a molecular test for Mycobacterium tuberculosis

SUMMARY:
The overall objective of this Aim is to design and iteratively adapt a home-based, mHealth- and oral testing facilitated strategy for implementing tuberculosis (TB) contact tracing in Cali, Colombia. Investigators will employ an iterative, community-engaged, participatory co-design process to optimize the feasibility, acceptability, usability, and appropriateness of the mobile health (mHealth) and oral testing strategy, in preparation for a future, appropriately powered implementation-effectiveness trial.

This protocol includes the baseline contact tracing protocol and the procedures for determining adaptations to the mHealth strategy (i.e., nominal group technique).

DETAILED DESCRIPTION:
This study will examine the diagnostic performance of oral samples for TB molecular testing in clinic and household settings; as well as utilize a community-engaged design methodology to iteratively refine a mHealth strategy for implementing contact tracing optimized for feasibility, acceptability, usability, and appropriateness.

There is a Certificate of Confidentiality in place for this study.

After contact tracing procedures have concluded, investigators will administer study instruments to characterize the feasibility, acceptability, appropriateness, and usability of the chatbot. Investigators will also conduct up to ~12 key informant interviews with purposively sampled index persons with TB and their household contacts to elicit views on the mHealth strategy during each cycle (for a total of up to ~36 key informant interviews).

After ~40 households (index persons with TB and their household contacts) have been enrolled using these procedures, and all scales and key informant interviews have been completed, the mHealth implementation strategy will be adapted using nominal group technique. Investigators will repeat this cycle twice for a total of three rounds of design and adaptation of chatbot-facilitated contact tracing procedures.

ELIGIBILITY:
Inclusion Criteria:

For index persons with TB:

* assigned by the SoPH to receive contact investigation services from the study community health worker
* may be of any age (represented by a parent or legal guardian for those age<18)

For contacts of index persons with TB:

* include the index person's named household contacts, defined as those spending one or more days or nights within the past 3 months sleeping under the same roof as the index person;
* may be of any age (represented by a parent or legal guardian for those age<18).

Exclusion Criteria:

For index persons with TB:

* who are living outside the city of Cali;
* who lack capacity to agree to testing.

For contacts of index persons with TB:

* who have already been diagnosed with and treated for active TB within the past two years;
* who lack capacity to agree to testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Lucian Davis, MD, Principal Investigator — Yale School of Public Health
Locations (1):
- Centro Internacional de Entrenamiento e Investigaciones Medicas (CIDIEM), Cali, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data arising from the project will be stored at Dryad, an online, open-access data repository.
Time Frame: The data will be made available immediately at the time of publication of the results. Data will be available for at least 5 years.
Access Criteria: Data will be searchable at the Dryad repository through keyword or through a unique identifier that will be published with the manuscript or made available on request of the corresponding author.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No randomization in this trial. Single arm interventional study.
Period: Overall Study
Arm/Group | Mobile Health and Oral Testing
Started | 269
Completed | 217
Not Completed | 52
Not completed — No intervention received due to inaccurate contact info, no WhatsApp, no internet, or no smartphone | 52

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Health and Oral Testing
Number analyzed (Participants) | 269
Age, Continuous [Median (Full Range); unit: years] | 43 [18 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 160
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Colombia | 269
Person living with HIV [Count of Participants; unit: Participants] — Only measured among those with tuberculosis (n=191) Population: Only measured among those with tuberculosis (n=191)
  Participants
    number analyzed (Participants) | 191
    (all) | 17
Pulmonary tuberculosis [Count of Participants; unit: Participants] — Only among those with tuberculosis (n=191) Population: Only among those with tuberculosis (n=191)
  Participants
    number analyzed (Participants) | 191
    (all) | 166
Person with tuberculosis [Count of Participants; unit: Participants] | 191
Contact of person with tuberculosis [Count of Participants; unit: Participants] | 78

OUTCOME MEASURES:

1. Primary Outcome: Implementation of the mHealth Strategy to Assess Feasibility.
Description: Feasibility of the mHealth strategy was defined as the proportion of index persons with TB and household contacts at risk of TB who engaged with the chatbot, defined as responding to at least one message from the chatbot.
Time Frame: within 14 days of invitation
Population: Number of individuals who successfully received the chatbot. 52 did not receive the chatbot. We did not collect reasons why the chatbot was not received.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health and Oral Testing
Number analyzed (Participants) | 217
Participants | 112

2. Primary Outcome: Oral Specimen Collection to Assess Feasibility.
Description: Feasibility of the oral testing strategy defined as the proportion of eligible and enrolled contacts of the index person with TB with successful collection of an oral sample
Time Frame: within 7 days of screening
Population: Investigators were unable to pilot the oral testing strategy within contacts of persons with tuberculosis as the Ministry of Health cancelled the contract with the community health workers. Without the community health workers in place, this strategy was infeasible and will not be collected in the future.
Arm/Group | Mobile Health and Oral Testing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not collected as part of this pilot as the chatbot was considered to be low risk to participant
Description: No definition of AEs
Arm/Group | Mobile Health and Oral Testing
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT06338462/Prot_000.pdf